CLINICAL TRIAL: NCT04347317
Title: Can High Intensity Inspiratory Muscle Training Improve Inspiratory Muscle Strength and Accelerate Weaning in Medical Patients With Difficulty on Weaning Admitted in the Intensive Care Unit?
Brief Title: Can High Intensity Inspiratory Muscle Training Improve Inspiratory Muscle Strength and Accelerate Weaning in Medical Patients With Difficulty on Weaning?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PR(ATR)03/2020
Record Dates: First submitted 2020-04-09; First posted 2020-04-15 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Weaning Failure
Keywords: mechanical ventilator weaning; mechanical ventilation; difficult weaning; intensive care unit; inspiratory muscle training; ventilator-induced diaphragmatic dysfunction; physiotherapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low Intensity IMT (Active Comparator)
  Interventions: Procedure: Low Intensity IMT
- High Intensity IMT (Experimental)
  Interventions: Procedure: High Intensity IMT

INTERVENTIONS:
Procedure: Low Intensity IMT — The control group will get a supervised IMT with Threshold IMT device, once a day, 5 days a week for a maximum of 28 days or until the participant is weaned successfully. In each session the participant will do 5 sets of 6 repetitions with 2 minutes of rest between sets. The initial training load will be adjusted to 30% of the MIP and will be increased by 10% of the initial MIP weekly.
  The patient will be placed in a semi-incorporated position (head of the bed elevated 45º). The ICU physiotherapist will check before training that the cuff of the tracheal tube is correctly swollen to avoid air leaks during the training. The ICU physiotherapist will disconnect the mechanical ventilation during the IMT and will provide supplemental oxygen when required. However, between series the participant will be returned to ventilator support. Patients will be instructed to do a whole expiration and immediately inspire as forceful as possible until reaching the total lung capacity.
  Arms: Low Intensity IMT
Procedure: High Intensity IMT — The experimental group will get a supervised IMT with Threshold IMT device, once a day, 5 days a week for a maximum of 28 days or until the participant is weaned successfully. In each session the participant will do 5 sets of 6 repetitions with 2 minutes of rest between sets. The initial training load will be adjusted to 60% of the MIP and will be increased by 10% of the initial MIP weekly.
  The patient will be placed in a semi-incorporated position (head of the bed elevated 45º). The ICU physiotherapist will check before training that the cuff of the tracheal tube is correctly swollen to avoid air leaks during the training. The ICU physiotherapist will disconnect the mechanical ventilation during the IMT and will provide supplemental oxygen when required. However, between series the participant will be returned to ventilator support. Patients will be instructed to do a whole expiration and immediately inspire as forceful as possible until reaching the total lung capacity.
  Arms: High Intensity IMT

SUMMARY:
Introduction: It has been described that invasive mechanical ventilation leads to diaphragm weakness. The inspiratory muscle weakness is related with a difficult and prolonged weaning as well as longer duration of mechanical ventilation and increased risk of complications and death. Consequently, the duration of stay in ICU is longer and the costs in ICU increase.

Objectives: To determine the effects of a high intensity inspiratory muscle training (IMT) on inspiratory muscle strength, weaning outcomes, complications and length of stay in the ICU in medical patients with difficulty on weaning and admitted in the ICU.

Methodology: In a single blind randomized clinical trial, 40 tracheotomy ventilated medical patients in which spontaneous breathing trial has failed ≥ 1 time, will be selected and randomized into two equitable groups. In the intervention group, IMT will be performed at 60% of the maximum inspiratory pressure (which will increase by 10% every week) while in the control group it will be performed at 30%. In both groups, 5 sets of 6 breaths will be performed, once a day, 5 days a week, for a maximum of 28 days or until the patient is successfully weaned. The main outcome will be the maximum inspiratory pressure, while the maximum expiratory pressure, weaning duration process, weaning success, duration of mechanical ventilation, length of stay in the ICU, complications and the rapid shallow breathing index will be analyzed as secondary outcomes.

t-student test for independent samples will be used to analyze quantitative outcomes. For qualitative outcomes will be used X2 test. A value of p<0.05 will be assumed as an indicator of statistically significant results.

Future contributions: Our collect results can be useful for the updating of the clinical practice guidelines and promote its implementation in the clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Medical patients aged ≥ 18 years hospitalized in the ICU.
* Patients ventilated by tracheostomy and who have failed ≥ 1 spontaneous breathing test.
* Being ventilated in assisted-controlled, assisted or pressure support modes.
* PEEP ≤ 10 cmH2O
* Richmond Agitation-Sedation Scale between -1 and 0.
* Confusion Assessment Method for the Intensive Care Unit negative.
* Cardiorespiratory and hemodynamic stability in the absence of vasopressor support or with minimal requirement (dobutamine or dopamine ≤ 5 μg / kg / min, phenylephrine ≤ 1 μg / kg / min).
* FiO2 ≤ 0,6
* PaO2/FiO2 ratio > 200
* Blood lactate levels < 4 mmol/L

Exclusion Criteria:

* Progressive neuromuscular disease
* Thoraco-abdominal surgery in a period <30 days from the beginning of the study.
* Diseases that cause hemodynamic instability (cardiac arrhythmia, decompensated heart failure, unstable ischemic heart disease).
* Hemoptysis
* Unstable chest wall.
* Not drained pneumothorax
* Phrenic nerve injury
* Spinal cord injury above T8
* Clinical signs of respiratory distress (paradoxal breathing, use of accessory respiratory muscles)
* Body mass index > 40 kg / m2
* Use domiciliary ventilator support prior to hospitalization.
* Skeletal disorder of the rib cage that impairs its biomechanics (severe kyphoscoliosis, congenital deformities).
* Body temperature > 38ºC
* Pregnancy
* Receive therapy with nitric oxide or nebulized prostacyclin.
* Medical order.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2021-09-15 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Inspiratory muscle strength | Through study completion, an average of 28 days
  Measured with MIP (Maximal Inspiratory Pressure)
  Assessments:
  Baseline, after the intervention period

SECONDARY OUTCOMES:
Expiratory muscle strength | Through study completion, an average of 28 days
  Measured with MEP (Maximal Expiratory Pressure)
  Baseline, after the intervention period
Rapid Shallow Breathing Index | Through study completion, an average of 28 days
  Measured with the mechanical ventilator
Duration of the weaning period | Through study completion, an average of 28 days
  Defined as the hours since the first attempt of spontaneous breathing (or the initiation of pressure support ≤ 7 cmH2O) to successful weaning
Weaning success | Through study completion, an average of 28 days
  Recorded as successfully if the patient can breathe spontaneously through tracheostomy without restart mechanical ventilation for at least 48 hours.
Duration of mechanical ventilation | Through study completion, an average of 28 days
  Recorded as the days since patient was connected to mechanical ventilator to successful weaning.
Length of stay in the ICU | Through study completion, an average of 28 days
  Measured in days.
Complications | Through study completion, an average of 28 days
  Defined as the patient needs to be intubated again when the patient was weaned or the death of the participant

CONTACTS AND LOCATIONS:
Overall Officials: Bernat Planas Pascual, PT,MSc, Principal Investigator — Hospital Universitari Vall d'Hebron Research Institute
Locations (2):
- Spain (2):
  - Hospital Universitari Vall d'Hebron Research Institute, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dixit A, Prakash S. Effects of threshold inspiratory muscle training versus conventional physiotherapy on the weaning period of mechanically ventilated patients: a comparative study. Int J Physiother Res. 2014;2(2):424-8
- [Background] Moodie L, Reeve J, Elkins M. Inspiratory muscle training increases inspiratory muscle strength in patients weaning from mechanical ventilation: a systematic review. J Physiother. 2011;57(4):213-21. doi: 10.1016/S1836-9553(11)70051-0. PMID 22093119
- [Background] Bonnevie T, Villiot-Danger JC, Gravier FE, Dupuis J, Prieur G, Medrinal C. Inspiratory muscle training is used in some intensive care units, but many training methods have uncertain efficacy: a survey of French physiotherapists. J Physiother. 2015 Oct;61(4):204-9. doi: 10.1016/j.jphys.2015.08.003. Epub 2015 Sep 11. PMID 26365266
- [Background] Bissett B, Leditschke IA, Green M, Marzano V, Collins S, Van Haren F. Inspiratory muscle training for intensive care patients: A multidisciplinary practical guide for clinicians. Aust Crit Care. 2019 May;32(3):249-255. doi: 10.1016/j.aucc.2018.06.001. Epub 2018 Jul 11. PMID 30007823
- [Background] Tonella RM, Ratti LDSR, Delazari LEB, Junior CF, Da Silva PL, Herran ARDS, Dos Santos Faez DC, Saad IAB, De Figueiredo LC, Moreno R, Dragosvac D, Falcao ALE. Inspiratory Muscle Training in the Intensive Care Unit: A New Perspective. J Clin Med Res. 2017 Nov;9(11):929-934. doi: 10.14740/jocmr3169w. Epub 2017 Oct 2. PMID 29038671
- [Background] Condessa RL, Brauner JS, Saul AL, Baptista M, Silva AC, Vieira SR. Inspiratory muscle training did not accelerate weaning from mechanical ventilation but did improve tidal volume and maximal respiratory pressures: a randomised trial. J Physiother. 2013 Jun;59(2):101-7. doi: 10.1016/S1836-9553(13)70162-0. PMID 23663795
- [Background] Bissett B, Leditschke IA, Green M. Specific inspiratory muscle training is safe in selected patients who are ventilator-dependent: a case series. Intensive Crit Care Nurs. 2012 Apr;28(2):98-104. doi: 10.1016/j.iccn.2012.01.003. Epub 2012 Feb 15. PMID 22340987
- [Background] Sassoon CS, Caiozzo VJ, Manka A, Sieck GC. Altered diaphragm contractile properties with controlled mechanical ventilation. J Appl Physiol (1985). 2002 Jun;92(6):2585-95. doi: 10.1152/japplphysiol.01213.2001. PMID 12015377
- [Background] Levine S, Nguyen T, Taylor N, Friscia ME, Budak MT, Rothenberg P, Zhu J, Sachdeva R, Sonnad S, Kaiser LR, Rubinstein NA, Powers SK, Shrager JB. Rapid disuse atrophy of diaphragm fibers in mechanically ventilated humans. N Engl J Med. 2008 Mar 27;358(13):1327-35. doi: 10.1056/NEJMoa070447. PMID 18367735
- [Background] Hudson MB, Smuder AJ, Nelson WB, Bruells CS, Levine S, Powers SK. Both high level pressure support ventilation and controlled mechanical ventilation induce diaphragm dysfunction and atrophy. Crit Care Med. 2012 Apr;40(4):1254-60. doi: 10.1097/CCM.0b013e31823c8cc9. PMID 22425820
- [Background] Silva PE. Inspiratory muscle training in mechanical ventilation: suitable protocols and endpoints, the key to clear results - a critical review. ASSOBRAFIR Ciência. 2015;6(1):21-30
- [Background] Elbouhy MS, AbdelHalim HA, Hashem AMA. Effect of respiratory muscles training in weaning of mechanically ventilated COPD patients. Egypt J Chest Dis Tuberc. 2014;63(3):679-87
- [Background] Bissett B, Leditschke IA. Inspiratory muscle training to enhance weaning from mechanical ventilation. Anaesth Intensive Care. 2007 Oct;35(5):776-9. doi: 10.1177/0310057X0703500520. PMID 17933168
- [Background] Sprague SS, Hopkins PD. Use of inspiratory strength training to wean six patients who were ventilator-dependent. Phys Ther. 2003 Feb;83(2):171-81. PMID 12564952
- [Background] Cader SA, Vale RG, Castro JC, Bacelar SC, Biehl C, Gomes MC, Cabrer WE, Dantas EH. Inspiratory muscle training improves maximal inspiratory pressure and may assist weaning in older intubated patients: a randomised trial. J Physiother. 2010;56(3):171-7. doi: 10.1016/s1836-9553(10)70022-9. PMID 20795923
- [Background] Hernández-López GH; Cerón-Juárez R; Escobar-Ortiz D; Graciano-Gaytán L; Gorordo-Delsol LA; Merinos-Sánchez G; Castañón-González JA; Amezcua-Gutiérrez MA; Cruz-Montesinos S; Garduño-López J; Lima-Lucero IM; Montoya-Rojo JO. Retiro de la ventilación mecánica. Med Crit. 2017;31(4):238-45
- [Background] Sandoval Moreno LM, Casas Quiroga IC, Wilches Luna EC, Garcia AF. Efficacy of respiratory muscle training in weaning of mechanical ventilation in patients with mechanical ventilation for 48hours or more: A Randomized Controlled Clinical Trial. Med Intensiva (Engl Ed). 2019 Mar;43(2):79-89. doi: 10.1016/j.medin.2017.11.010. Epub 2018 Feb 3. English, Spanish. PMID 29398169
- [Background] Medrinal C, Prieur G, Frenoy E, Robledo Quesada A, Poncet A, Bonnevie T, Gravier FE, Lamia B, Contal O. Respiratory weakness after mechanical ventilation is associated with one-year mortality - a prospective study. Crit Care. 2016 Jul 31;20(1):231. doi: 10.1186/s13054-016-1418-y. PMID 27475524
- [Background] Martin AD, Davenport PD, Franceschi AC, Harman E. Use of inspiratory muscle strength training to facilitate ventilator weaning: a series of 10 consecutive patients. Chest. 2002 Jul;122(1):192-6. doi: 10.1378/chest.122.1.192. PMID 12114357
- [Background] Vorona S, Sabatini U, Al-Maqbali S, Bertoni M, Dres M, Bissett B, Van Haren F, Martin AD, Urrea C, Brace D, Parotto M, Herridge MS, Adhikari NKJ, Fan E, Melo LT, Reid WD, Brochard LJ, Ferguson ND, Goligher EC. Inspiratory Muscle Rehabilitation in Critically Ill Adults. A Systematic Review and Meta-Analysis. Ann Am Thorac Soc. 2018 Jun;15(6):735-744. doi: 10.1513/AnnalsATS.201712-961OC. PMID 29584447
- [Background] Caruso P, Denari SD, Ruiz SA, Bernal KG, Manfrin GM, Friedrich C, Deheinzelin D. Inspiratory muscle training is ineffective in mechanically ventilated critically ill patients. Clinics (Sao Paulo). 2005 Dec;60(6):479-84. doi: 10.1590/s1807-59322005000600009. Epub 2005 Dec 12. PMID 16358138
- [Background] Mohamed AR, El Basiouny HMS, Salem NM. Response of Mechanically Ventilated Respiratory Failure Patients to Respiratory Muscles Training. Med J Cairo Univ. 2014;82(1):19-24
- [Background] Ibrahiem AA;, Mohamed AR;, Saber HM; Effect Of Respiratory Muscles Training In Addition To Standard Chest Physiotherapy On Mechanically Ventilated Patients. J Med Res Pract. 2014;3(3):52-8
- [Background] Martin AD, Smith BK, Davenport PD, Harman E, Gonzalez-Rothi RJ, Baz M, Layon AJ, Banner MJ, Caruso LJ, Deoghare H, Huang TT, Gabrielli A. Inspiratory muscle strength training improves weaning outcome in failure to wean patients: a randomized trial. Crit Care. 2011;15(2):R84. doi: 10.1186/cc10081. Epub 2011 Mar 7. PMID 21385346
- [Background] Downey AE, Chenoweth LM, Townsend DK, Ranum JD, Ferguson CS, Harms CA. Effects of inspiratory muscle training on exercise responses in normoxia and hypoxia. Respir Physiol Neurobiol. 2007 May 14;156(2):137-46. doi: 10.1016/j.resp.2006.08.006. Epub 2006 Sep 22. PMID 16996322
- [Background] Girard TD, Alhazzani W, Kress JP, Ouellette DR, Schmidt GA, Truwit JD, Burns SM, Epstein SK, Esteban A, Fan E, Ferrer M, Fraser GL, Gong MN, Hough CL, Mehta S, Nanchal R, Patel S, Pawlik AJ, Schweickert WD, Sessler CN, Strom T, Wilson KC, Morris PE; ATS/CHEST Ad Hoc Committee on Liberation from Mechanical Ventilation in Adults. An Official American Thoracic Society/American College of Chest Physicians Clinical Practice Guideline: Liberation from Mechanical Ventilation in Critically Ill Adults. Rehabilitation Protocols, Ventilator Liberation Protocols, and Cuff Leak Tests. Am J Respir Crit Care Med. 2017 Jan 1;195(1):120-133. doi: 10.1164/rccm.201610-2075ST. PMID 27762595